CLINICAL TRIAL: NCT04160052
Title: Phase I/II of Venetoclax in Combination With Azacitidine in Treatment Naïve and Relapse Refractory High Risk MDS Individuals"
Brief Title: Venetoclax and Azacitidine for the Treatment of High-Risk Recurrent or Refractory Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0368; NCI-2019-06873 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0368 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-04; First posted 2019-11-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Recurrent Myelodysplastic Syndrome; Refractory Myelodysplastic Syndrome; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, azacitidine) (Experimental): Patients receive venetoclax orally PO QD on days 1-7 or 1-14 and azacitidine SC or IV over 15 minutes on days 1-5. Cycles repeat every 4-8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I/II trial studies the side effects and best dose of venetoclax when given together with azacitidine in treating patients with high-risk myelodysplastic syndrome that has come back (recurrent) or does not respond to treatment (refractory). Drugs used in chemotherapy, such as venetoclax and azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability (phase 1) and overall response rate (ORR) (phase 2) of venetoclax in combination with azacitidine in patients with treatment-naive high-risk myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) with bone marrow excess blasts > 5% and patients that are relapsed/refractory to prior hypomethylating agent (HMA) therapy.

SECONDARY OBJECTIVES:

I. Rate of complete remission (CR). II. Rate of marrow/morphologic complete remission (mCR). III. Rate of hematologic improvement (HI; erythroid/platelet/neutrophil responses).

IV. Rate of red blood cell (RBC) transfusion independence. V. Rate of platelet (PLT) transfusion independence. VI. Rate of cytogenetic response. VII. Rate of bone marrow blast response. VIII. Time to transformation to acute myeloid leukemia (AML). IX. Duration of response (DOR). X. Overall survival (OS). XI. Progression-free survival (PFS). XII. Time to next MDS treatment (TTNT). XIII. Event-free survival (EFS).

EXPLORATORY OBJECTIVE:

I. To investigate the effects of therapy on MDS and to identify biological markers of response to venetoclax and/or its combination with azacitidine.

OUTLINE: This is a phase I, dose-escalation study of venetoclax followed by a phase II study.

Patients receive venetoclax orally (PO) once daily (QD) on days 1-7 or 1-14 and azacitidine subcutaneously (SC) or intravenously (IV) over 15 minutes on days 1-5. Cycles repeat every 4-8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* For phase I, patients can be HMA-naive high-risk MDS (Int-2 or high risk by the International Prognostic Scoring System [IPSS] with overall score >= 1.5) with excess blasts > 5%, or relapsed/refractory MDS post-HMA failure (defined as prior receipt of 4 cycles of HMA therapy with failure to attain a response, or progression of disease or relapse at any time after prior response to HMA therapy) with > 5% blasts
* For phase II, patients will be divided into 2 cohorts: Cohort A: patients with HMA-naive high-risk MDS (Int-2 or high risk by the IPSS with overall score >= 1.5) with excess blasts > 5%. Cohort B: patients with relapsed/refractory MDS post-HMA failure (defined as prior receipt of 4 cycles of HMA therapy with failure to attain a response, or progression of disease or relapse at any time after prior response to HMA therapy) with > 5% blasts are eligible. Note: Patients with chronic myelomonocytic leukemia (CMML) and therapy-related MDS are eligible. Hydroxyurea is allowed to lower the white cell count =< 10,000/ul prior to initiation of venetoclax
* Total bilirubin < 3 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Alanine aminotransferase (ALT) < 4 x ULN unless considered due to leukemic involvement
* Creatinine < 2 x ULN unless related to the disease
* Signed written informed consent. Consent may be translated for Non-English Speaking Patients per institutional policy.
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment
* Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment

Exclusion Criteria:

* Patients having received any prior BCL2 inhibitor therapy
* Patients with MDS with IPSS risk categories low or Int-1 (overall IPSS score < 1.5)
* Pregnant or breastfeeding
* Cognitively impaired patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-02-03 (Actual); Study Completion 2026-02-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of the combination regimen of venetoclax and azacitidine (Phase I) | Up to 8 weeks
  The MTD is the highest dose level in which < 2 patients of 6 develop first cycle dose-limiting toxicity.
Incidence of adverse events (Phase I) | Up to 5 years
  Safety data will be summarized by category, severity, and frequency.

SECONDARY OUTCOMES:
Overall response rate (Phase 2) | Up to 5 years
  Will be defined as the proportion of patients who had complete remission (CR), partial remission (PR), marrow complete remission, or hematologic improvement lasting at least 4 weeks. Will estimate the overall response rate for the combination treatment, along with the 95% confidence interval.
Rate of CR | Up to 5 years
  The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Rate of marrow/morphologic CR | Up to 5 years
  The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Rate of hematologic improvement | Up to 5 years
  The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Rate of red blood cell transfusion independence | Up to 5 years
Rate of platelet transfusion independence | Up to 5 years
  The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Rate of cytogenetic response | Up to 5 years
  The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Rate of bone marrow blast response | Up to 5 years
  The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Time to transformation to acute myeloid leukemia | Up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Duration of response | From the date of initial response (PR or better) to the date of first documented disease progression/relapse or death, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Overall survival | From treatment start till death or last follow-up, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Progression-free survival | From treatment to progression or last follow-up, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Time to next myelodysplastic syndrome treatment | Up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Event-free survival | From the date of treatment initiation to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.

OTHER OUTCOMES:
Effects of therapy on myelodysplastic syndrome | Up to 5 years
Biological markers of response | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bazinet A, Darbaniyan F, Jabbour E, Montalban-Bravo G, Ohanian M, Chien K, Kadia T, Takahashi K, Masarova L, Short N, Alvarado Y, Yilmaz M, Ravandi F, Andreeff M, Kanagal-Shamanna R, Ganan-Gomez I, Colla S, Qiao W, Huang X, McCue D, Mirabella B, Kantarjian H, Garcia-Manero G. Azacitidine plus venetoclax in patients with high-risk myelodysplastic syndromes or chronic myelomonocytic leukaemia: phase 1 results of a single-centre, dose-escalation, dose-expansion, phase 1-2 study. Lancet Haematol. 2022 Oct;9(10):e756-e765. doi: 10.1016/S2352-3026(22)00216-2. Epub 2022 Sep 2. PMID 36063832
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT04160052/ICF_000.pdf